CLINICAL TRIAL: NCT04306770
Title: Optimizing Care of Patients Via Telehealth In Monitoring and Augmenting Their Control of Diabetes Mellitus
Acronym: OPTIMUM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SingHealth Polyclinics (Other)
Collaborators: MOH Office for Healthcare Transformation (MOHT), Singapore (Unknown); Phillips Healthcare, Singapore (Unknown); Reinsurance Group of America (RGA), Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019/2340
Record Dates: First submitted 2020-03-06; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): OPTIMUM Programme
  Interventions: Other: OPTIMUM programme
- Control (No Intervention): Treatment as usual

INTERVENTIONS:
Other: OPTIMUM programme — OPTIMUM programme encompass of telehealth service to support the patient. Study participants will be given devices (Bluetooth-enabled blood pressure machine, weighing scale and glucometer) to monitor their parameters at home. Care team will use the Phillips "Vital Health" to perform tele-monitoring, tele-management (individualized on-line health coaching and timely interventions), and to deliver education content.
  Arms: Intervention

SUMMARY:
OPTIMUM study aims to use the telehealth-enabled chronic disease management programme for individuals with chronic diseases to provide timely intervention to prevent disease deterioration, increase compliance to treatment regimen (e.g. medication), and most importantly, engage participants to better manage their own care.

DETAILED DESCRIPTION:
Over 400,000 Singaporeans are living with diabetes, with PM Lee Hsien Loong calling it a "health crisis" and the Ministry of Health declaring a "War on Diabetes" in 2016. One in three Singaporeans has a lifetime risk of getting diabetes and the number of those with diabetes is projected to reach one million by 2050, if current trends continue. Life years lost due to mortality and ill-health related to diabetes was the 4th largest among all diseases in 2010 while the cost burden from diabetes, including medical expenses and productivity loss, was expected to rise from beyond $940 million in 2014 to $1.8 billion in 2050. In addition, every year in Singapore, 2 in 3 new kidney failure cases are due to diabetes, and 1 in 2 people who suffer from a heart attack had co-existing diabetes. Tele-health projects have been conducted successfully overseas on patients suffering from diabetes.

Telehealth refers to the systematic provision of healthcare services over physically separate environments via Information and Communications Technology (ICT) and distinguishes between four main dimensions/ domains of Telemedicine as follow:

1. Tele-collaboration, which refers to interactions between (facility-based or mobile) onsite and remote healthcare professionals for clinical purposes e.g. referral, co-diagnosis, supervision or case review. The distinguishing feature is that healthcare professionals are involved at both ends of the interaction and a patient may or may not be involved in the same Telemedicine interaction.
2. Tele-treatment, which refers to interactions between remote healthcare professionals and patients/ caregivers for the purposes of direct clinical care. The distinguishing feature is that a patient or caregiver is involved directly at one end of the interaction and this creates (or presupposes the existence of) a professional-patient relationship. Tele-treatment is used in the remote delivery of primary care and many forms of speciality care.
3. Tele-monitoring, which refers to biomedical and other forms of data collection directly from patients (or through caregivers) by remote systems, which are used by healthcare professionals for clinical purposes such as vital signs monitoring and home nursing. Tele-monitoring is used in remote chronic disease management. The distinguishing feature is that a healthcare professional or organisation is engaged at one end. Another feature of Tele-monitoring is that it need not create (or presuppose the existence of) a professional-patient relationship even though the healthcare organisation as a whole might ow a duty of care to the patient.
4. Tele-support, which refers to the use of online services for non-clinical (ie educational and administrative) purposes to support the patient, and caregiver. The "More Independent" programme run by Philips and the Liverpool Clinical Commissioning Group (CCG) provided telehealth services for 1,808 patients recruited from the primary care setting in Liverpool. The study showed reductions in emergency admissions and secondary care costs (in comparison with the control group) ranging from 22% to 32% for patients with above average risk (25% or more). Patient reported outcomes (PRO) also show that 90% of patients feel more in control, have gained confidence and/or feel better able to cope with their condition.

However, there has been no such large scale study done in Singapore to study the impact of telehealth on the disease progression, healthcare utilisation and cost of care for diabetic patients in the primary care setting. As such, an evaluation of a prospective telehealth programme, i.e. Optimizing care of Patients via Telehealth In Monitoring and Augmenting their control of Diabetes Mellitus (OPTIMUM) is being planned for in SingHealth Polyclinics.

The current standard of care comprises on-site measurements of clinical parameters and education in a usual outpatient clinic setting. The telehealth programme comprises remote patient monitoring, education, individualised on-line health coaching and timely interventions provided by primary healthcare professionals in polyclinics. The proposed Philips VitalHealth solution incorporates telehealth-enabled chronic disease management and care coordination. The telehealth-enabled chronic disease management programme is customised for individuals with chronic diseases and aims to provide timely intervention to prevent disease deterioration, increase compliance to treatment regimen (e.g. medication), and most importantly, engage participants to better manage their own care.

On the insurance front, there are many "gaps" present in the insurance industry today with regard to chronic diseases, and to this end, Reinsurance Group of America (RGA) is interested to jointly study the effectiveness of a telehealth programme on diabetic patients, so that they can develop new health insurance products that can meet that insurance gap.

ELIGIBILITY:
Inclusion Criteria:

1 . Singapore Citizen or Permanent Resident

2. Age 26 - 65 years (latest age of entry for insurance coverage is 65 at next birthday)

3. Type 2 Diabetes Mellitus (HbA1c ≤ 10% and ≥ 7.5% per latest reading) with and without the following complications:

1. Mild non-proliferative diabetic retinopathy without any macular or retinal involvement;
2. Chronic Kidney Diseases up to stage 3

   4. Patients registered with participating polyclinic

   5. Non-smoker, or ex-smoker who has completely quit smoking for at least 12 months

   6. Existing user of smartphone and is willing to download the relevant mobile application (iPhone or Android phones are acceptable)

   7. Expressed willingness to use the telehealth system and devices according to study protocol during the study period

Exclusion Criteria:

1. Poorly controlled glycemic control with HbA1c > 10% (latest reading)
2. Cognitively impaired based on diagnosis of dementia or mild cognitive impairment (MCI) in the electronic health records (EHR)
3. Existing conditions listed below, as documented in the EHR:

   1. Any proliferative diabetic retinopathy (moderate to severe) and any macular or other retinal complications;
   2. Chronic kidney disease Stage 4 or 5;
   3. Coronary arterial diseases.
   4. Cerebrovascular diseases such as transient ischemic attach (TIA) or stroke;
   5. Peripheral vascular disease (result from diabetic foot screening);
   6. Known cognitive impairment, including MCI
4. Not able to use smartphone despite coaching
5. Any end-stage disease with life prognosis of < 2 year
6. Patients who are not willing or are not able to commit to the entire Optimum program
7. Pregnant women
8. Currently enrolled in another study / programme involving a novel therapeutic drug or device

Ages: 26 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Diabetic control | 6 months
  HbA1c (in percentage)

SECONDARY OUTCOMES:
Diabetic control | 12 months, 24 months
  HbA1c (in percentage)
Blood pressure control | 6 months, 12 months, 24 months
  Systolic and diastolic blood pressure (in mmHg)
Optimal weight control | 6 months, 12 months, 24 months
  Weight (in kilogram)
Utility Score | 6 months, 12 months, 24 months
  EQ-5D-5L questionnaire, reported as index value by applying the formula. the higher the score the better.
  * EQ-5D-5L is not an abbreviation
Diabetic medication adherence 9 Diabetic medication adherence (Oral Hypoglycemia agent) | 6 months, 12 months, 24 months
  Medication Adherence Rating Scale 5 (MARS 5) - max score of 25, min score of 5 (the higher the score the better the adherence)
Diabetic medication adherence (Insulin) | 6 months, 12 months, 24 months
  Medication possession ratio (MPR) - max score of 1, min score of 0, higher number indicate better adherence
Diabetic knowledge | 6 months, 12 months, 24 months
  23 items Michigan Diabetes Research and Training Center's revised Diabetes Knowledge Test - Max Score of 23, Min score of 0, the higher the score the better the knowledge
Diabetic self-care | 6 months, 12 months, 24 months
  Self-Care Inventory-Revised Version (SCI-R) scale- Max sore of 15, min score of 15 - the higher the score the better the self-care
Diabetes distress survey | 6 months, 12 months, 24 months
  Problem Areas in Diabetes Scale (PAID), Max score of 80, min score of 0, the lower the core the better (lesser distress)
Healthcare utilization | 6 months, 12 months, 24 months
  Healthcare cost
Incidence of vascular complications | 6 months, 12 months, 24 months
  Incidence of both micro- and macro- vascular complication

CONTACTS AND LOCATIONS:
Overall Officials: Ngiap Chuan Tan, FCFPS, Principal Investigator — SingHealth Polyclinics
Locations (1):
- Sengkang Polyclinic, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berkel C van, Smith M, Horsfield D, McManus H. Evidence for Supported Self-Care at Scale. International Journal of Integrated Care. 2016 Nov 9;16(5):S44.
- [Derived] Tan NC, Gong PP, Lee CS, Goh SKL, Ang SB, Koh GCH. Theory-based behaviour modification of Asian adults with type-2 diabetes mellitus after participating in a novel telemonitoring system: a qualitative research study. BMJ Open. 2024 Dec 23;14(12):e080830. doi: 10.1136/bmjopen-2023-080830. PMID 39719282
- [Derived] Goh KLS, Lee CS, Koh CHG, Ling NL, Ang SB, Oh C, Lin Y, Yuan W, Zheng QC, Tan NC. Evaluating the effectiveness and utility of a novel culturally-adapted telemonitoring system in improving the glycaemic control of Asians with type-2 diabetes mellitus: a mixed method study protocol. Trials. 2021 Apr 26;22(1):305. doi: 10.1186/s13063-021-05240-6. PMID 33902656
- See also: News higlight on Singapore goverment initiative in tackling diabetes. — https://www.moh.gov.sg/news-highlights/details/diabetes-the-war-continues
- See also: Report on the Singapore Burden of Diseases Study 2010 — https://policy.nl.go.kr/cmmn/FileDown.do?atchFileId=107157&fileSn=2883